CLINICAL TRIAL: NCT06838260
Title: Assessment of the Effects of Endotracheal Tube Temperature on Respiratory Complications in Children Undergoing Adenotonsillectomy
Brief Title: Assessment of Endotracheal Tube Temperature Effects in Children Undergoing Adenotonsillectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Mursel Ekinci, Assoc Prof, Bursa City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Bursa City Hospital 11
Record Dates: First submitted 2024-11-11; First posted 2025-02-20 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Adenotonsillectomy
Keywords: Adenotonsillectomy in children; Endotracheal tube temperature; Respiratory complications

STUDY DESIGN:
Intervention Model Description: There are two models for this study. Children intubated with an endotracheal tube which 24° celcius (Group T24), Children intubated with an endotracheal tube which 37° celcius (Group T37)
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and the outcomes assessor will not know the groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group T24 (24°C Endotracheal tube) (Active Comparator): Anesthesiologist will administer 0.02 mg/kg midazolam (Demizolam ®) for premedication 30 minutes before entering the operating room. The operating room temperature will be kept at 24°C. After entering the operating room, 1 mg/kg lidocaine (Aritmal ®), 2 mg/kg propofol (Propofol ®), 1 mcg/kg fentanyl (Fentanyl ®), 0.5 mg/kg rocuronium (Muscoblok ®) will be administered within the standard anesthesia induction protocol and the patients will be intubated by the anesthesiologist with age-appropriate endotracheal tube. After confirming the ETT location, the anesthesia device will be adjusted with age-appropriate respiratory rate and 6 l/kg tidal volume. Sevoflurane inhalation will be administered as 1 MAC for anesthesia maintenance. 10 mg/kg paracetamol will be administered to all patients for postoperative analgesia and 100 μg/kg Ondansetron for postoperative nausea and vomiting. At the end of surgery, 2mg/kg sugammadex will be administered for extubation.
  Interventions: Other: 24°C Endotracheal tube
- Group T37 (37°C Endotracheal tube) (Active Comparator): Anesthesiologist will administer 0.02 mg/kg midazolam (Demizolam ®) for premedication 30 minutes before entering the operating room. The operating room temperature will be kept at 24°C. After entering the operating room, 1 mg/kg lidocaine (Aritmal ®), 2 mg/kg propofol (Propofol ®), 1 mcg/kg fentanyl (Fentanyl ®), 0.5 mg/kg rocuronium (Muscoblok ®) will be administered within the standard anesthesia induction protocol and the patients will be intubated by the anesthesiologist with age-appropriate endotracheal tube. After confirming the ETT location, the anesthesia device will be adjusted with age-appropriate respiratory rate and 6 l/kg tidal volume. Sevoflurane inhalation will be administered as 1 MAC for anesthesia maintenance. 10 mg/kg paracetamol will be administered to all patients for postoperative analgesia and 100 μg/kg Ondansetron for postoperative nausea and vomiting. At the end of surgery, 2mg/kg sugammadex will be administered for extubation.
  Interventions: Other: 37°C Endotracheal tube

INTERVENTIONS:
Other: 24°C Endotracheal tube — A disposable ETT sized appropriately for the age of the patients will be kept in a 40°C incubator (MIR-162) for 30 minutes. An infrared non-contact thermometer will be used to measure the ETT wall temperature. After removal from the incubator, intubation will be performed as soon as the tubes reach a temperature of 24°C for the T1 group by serial measurements. All intubations will be performed by a single anesthesiologist who is not associated with the study.
  Arms: Group T24 (24°C Endotracheal tube)
Other: 37°C Endotracheal tube — A disposable ETT sized appropriately for the age of the patients will be kept in a 40°C incubator (MIR-162) for 30 minutes. An infrared non-contact thermometer will be used to measure the ETT wall temperature. After removal from the incubator, intubation will be performed as soon as the tubes reach a temperature of 37°C for the T2 group by serial measurements. All intubations will be performed by a single anesthesiologist who is not associated with the study.
  Arms: Group T37 (37°C Endotracheal tube)

SUMMARY:
Adenotonsillectomy is one of the most commonly performed surgical procedures in children worldwide. life-threatening complications such as laryngospasm and bronchospasm may develop in the postoperative period.

The aim of this study was to compare the effects of using endotracheal intubation tubes at different temperatures during intubation on respiratory complications in the postoperative period in children undergoing adenotonsillectomy.

DETAILED DESCRIPTION:
Adenotonsillectomy (AT) is one of the most common surgical procedures performed in children. Its incidence has been increasing day by day and has almost doubled since the 1970s. In recent years, with the development of surgical techniques and anesthetic approaches, significant progress has been made in the recovery and postoperative management of these patients and morbidity has decreased significantly. The most feared complications of AT in children are respiratuar complications such as laryngospasm and bronchospasm. These complications can occur during AT or in the postoperative period, requiring rapid response by the anesthesia and surgical team and extensive postoperative monitoring. They may result in increased morbidity and prolonged hospitalization. Different methods including intravenous lidocaine, topical lidocaine, propofol, iv magnesium and the like have been proposed to reduce laryngospasm; different results have been obtained in studies. Thermal softening of endotracheal tubes (ETT) with normal warm saline before intubation has been shown to be significantly effective in reducing sore throat and hoarseness during recovery and postoperatively. The aim of this study was to compare the intraoperative and postoperative respiratory effects of using endotracheal intubation tubes at different temperatures during intubation in children undergoing adenotonsillectomy.

ELIGIBILITY:
Inclusion Criteria:

* Parents who agreed to participate in the study
* Children undergoing adenotonsillectomy
* ASA 1 and 2 class patients

Exclusion Criteria:

* Emergency surgery
* Children with a history of difficult airway
* Children who have had upper airway surgery
* Presence or suspicion of upper or lower respiratory tract infection
* History of cardiac and respiratory diseases
* Patients with craniofacial malformations

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2025-03-02 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Rate of laryngospasm | From extubation until postoperative 2. hour
  The rates of laryngospasm occurring in the participants will be determined and compared between the 2 groups
Rate of bronchospasm | From extubation until postoperative 2. hour
  The rates of bronchospasm occurring in the participants will be determined and compared between the 2 groups
Rate of desaturation | From extubation until postoperative 2. hour
  The rates of desaturation occurring in the participants will be determined and compared between the 2 groups

SECONDARY OUTCOMES:
Heart rate | 7 times (1 minute(min) before induction of anaesthesia, 5 seconds(sec) after intubation, 5 min and 15 min after the start of surgery, 5 sec after the completion of surgery, 5 sec after extubation, 5 sec before transfer to post-anaesthesia care)
  Heart rate (HR) (bpm) will be recorded and data will be compared between groups
Mean arterial pressure (MAP) mmHg | 7 times (1 minute(min) before induction of anaesthesia, 5 seconds(sec) after intubation, 5 min and 15 min after the start of surgery, 5 sec after the completion of surgery, 5 sec after extubation, 5 sec before transfer to post-anaesthesia care)
  Mean arterial pressure (MAP) (mmHg) will be recorded and data will be compared between groups
Oxygen saturation | 7 times (1 minute(min) before induction of anaesthesia, 5 seconds(sec) after intubation, 5 min and 15 min after the start of surgery, 5 sec after the completion of surgery, 5 sec after extubation, 5 sec before transfer to post-anaesthesia care)
  Oxygen saturation (SpO2), (%) will be recorded and data will be compared between groups
Intraopearative anaesthesia machine respiratory data | 4 times measurement (5 seconds after intubation, 5 minutes after the start of surgery, 15 minutes after the start of surgery, 5 seconds after the completion of surgery)
  End-tidal carbon dioxide (EtCO2) (mmHg) will be recorded and data will be compared between groups
Intraopearative anaesthesia machine respiratory data 2 | 4 times measurement (5 seconds after intubation, 5 minutes after the start of surgery, 15 minutes after the start of surgery, 5 seconds after the completion of surgery)
  Maximum pressure measured at end inspiration (Ppeak) will be recorded and data will be compared between groups Mean airway pressure (Pmean) will be recorded and data will be compared between groups

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa City Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The investigators will not share IPD

REFERENCES:
- [Background] Jeyakumar A, Fettman N, Armbrecht ES, Mitchell R. A systematic review of adenotonsillectomy as a risk factor for childhood obesity. Otolaryngol Head Neck Surg. 2011 Feb;144(2):154-8. doi: 10.1177/0194599810392328. PMID 21634056
- [Background] Orestes MI, Lander L, Verghese S, Shah RK. Incidence of laryngospasm and bronchospasm in pediatric adenotonsillectomy. Laryngoscope. 2012 Feb;122(2):425-8. doi: 10.1002/lary.22423. Epub 2012 Jan 17. PMID 22252947
- [Background] Marzban S, Haddadi S, Naghipour MR, Sayah Varg Z, Naderi Nabi B. The effect of intravenous magnesium sulfate on laryngospasm after elective adenotonsillectomy surgery in children. Anesth Pain Med. 2014 Feb 28;4(1):e15960. doi: 10.5812/aapm.15960. eCollection 2014 Feb. PMID 24660159
- [Background] Mohseni M, Farahmand Rad R, Jafarian AA, Zarisfi AH, Masoudi N. The Effect of Softening of Endotracheal Tubes on the Decrement of Postoperative Hoarseness and Sore Throat. Anesth Pain Med. 2022 Nov 15;12(5):e123910. doi: 10.5812/aapm-123910. eCollection 2022 Oct. PMID 36937172
- [Background] Yu Y, Jia Q, Zhou L, Liu Z, Liang S, Yang Z, Wan Q. Appropriate tube temperature for fiberoptic bronchoscope-guided intubation of thermally softened double-lumen endotracheal tubes: A CONSORT-compliant article. Medicine (Baltimore). 2022 Oct 7;101(40):e29999. doi: 10.1097/MD.0000000000029999. PMID 36221346
- [Background] Komasawa N, Nishihara I, Tatsumi S, Minami T. Prewarming of the i-gel facilitates successful insertion and ventilation efficacy with muscle relaxation: a randomized study. J Clin Anesth. 2014 Dec;26(8):663-7. doi: 10.1016/j.jclinane.2014.08.009. Epub 2014 Nov 18. PMID 25468575